CLINICAL TRIAL: NCT05372861
Title: Nanopore Sequencing in Ophthalmology - a Paradigm Shift in Pathogen Determination?
Brief Title: Nanopore Sequencing in Ophthalmology
Status: Recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: NSIO
Record Dates: First submitted 2022-04-22; First posted 2022-05-13 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Endophthalmitis
Keywords: Endophthalmitis; Nanopore sequencing; Next Generation Sequencing
MeSH Terms: conditions — Endophthalmitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Vitreous and aqueous humor samples in eyes with endophthalmitis gathered during vitrectomy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this pilot study, the feasibility of the Oxford Nanopore MinION to identify pathogens from vitrectomy samples in eyes with endophthalmitis shall be assessed. The MinION is a low cost commercially available device for DNA/ RNA analysis that, in studies, has been used for pathogen determination in various infectious diseases as well as for the genetic characterization of hematologic tumors.

DETAILED DESCRIPTION:
Vitreous samples and anterior chamber taps from eyes with endophthalmitis are taken during routine vitrectomy. The gathered samples are divided in half to undergo routine culture for microbial growth and nanopore sequencing with the MinION Mk1b, a commercially available device for DNA/RNA sequencing. Base reads from Nanopore sequencing are then compared with available libraries for pathogen identification. The Nanopore sequencing results for pathogens are compared versus the results of the microbiological culture of the same eye as the gold standard. Clinical features and visual function before and after vitrectomy are gathered from patient charts. Treatment is not altered due to results of the Nanopore sequencing.

ELIGIBILITY:
Inclusion Criteria:

* Eyes of patients with endophthalmitis

Exclusion Criteria:

* No informed consent possible
* Participation in other studies

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Eyes of adult patients with endophthalmitis
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-04-22 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Pathogen detection | In vitro analysis after vitrectomy for endophthalmitis. Start of analysis: Within the next working day after sample acquisition. Time for Nanopore sequencing: Approximately up to 10 hours. Time for culture: 24 hours up to 14 days.
  Pathogens detected by Nanopore sequencing versus microbiologic culture

SECONDARY OUTCOMES:
Time to pathogen detection | Time measured from start of analysis until arrival of results. Time for Nanopore sequencing: Approximately up to 10 hours. Time for culture: 24 hours up to 14 days.
  Time in days from gathering of the sample until arrival of results
Visual acuity | Gathered from patient charts two months after vitrectomy.
  Visual acuity measured with Snellen charts

CONTACTS AND LOCATIONS:
Locations (1):
- Universitäts Augenklinik Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No